CLINICAL TRIAL: NCT02895503
Title: The Effect of Yoga and Exercise on the Quality of Life of Patients With Non-Small Cell Lung Cancer
Brief Title: Yoga in Improving Quality of Life in Patients With Non-small Cell Lung Cancer Undergoing Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual/Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-13850; NCI-2015-01818 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Non-small Cell Lung Cancer; Recurrent Non-Small Cell Lung Carcinoma
Keywords: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Yoga; Respiratory Physiological Phenomena; Vital Capacity; Peak Expiratory Flow Rate; Forced Expiratory Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (yoga) (Experimental): Patients undergo traditional medical treatment, participate in yoga comprising basic postures and breathing exercises 3-4 times per week, and attend yoga class once weekly over 30-60 minutes for 12 weeks.
  Interventions: Behavioral: Yoga; Other: FACT-L; Other: Pulmonary function test
- Arm II (emotional support group therapy) (Active Comparator): Patients undergo traditional medical treatment and participate in emotional support group therapy with a chaplain to work on mind-body therapies comprising guided imagery and spirituality once weekly for 12 weeks.
  Interventions: Behavioral: Support Group Therapy; Other: FACT-L; Other: Pulmonary function test

INTERVENTIONS:
Behavioral: Yoga — Participate in yoga
  Other Names: Yoga Therapy
  Arms: Arm I (yoga)
Behavioral: Support Group Therapy — Participate in emotional support group therapy
  Arms: Arm II (emotional support group therapy)
Other: FACT-L — This is a 44-item self-report instrument which measures multidimensional HRQOL. There are 5 sections dealing with physical, family, emotional, and functional well-being and their relationship with the doctor. There are nine questions in a sixth subscale that are specific to lung cancer (LSC), including shortness of breath, cough, etc. The TOI is the sum of the scores on the LCS and the physical well-being and functional well-being subscales of the FACT-L scale. The FACT-L has been shown to be reliable and valid and sensitive. (Cella, Bonomi, Lloyd, DS, Kaplan, & Bonomi, 1995). The instrument has been used with patients with lung cancer in the Massey Cancer Center.
  Other Names: Functional Assessment of Cancer Therapy - Lung
Other: Pulmonary function test — The pulmonary function test includes forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and peak expiratory flow rate (PEFR). Use of a digital spirometer provides an objective and reliable measure of the patient's vital capacity.
  Other Names: FVC, FEV1, PEFR; forced vital capacity, forced expiratory volume in 1 second, peak expiratory flow rate

SUMMARY:
The purpose of this research study is to evaluate the effects of yoga (including breathing exercises) on the quality of life in patients, diagnosed and undergoing standard treatments for non-small cell lung cancer.

DETAILED DESCRIPTION:
This clinical trial studies yoga in improving quality of life in patients with non-small cell lung cancer undergoing treatment. Yoga may help improve quality of life and pulmonary functional capacity in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any type of non-small cell lung cancer who are undergoing medical treatment, including surgery, radiation and / or chemotherapy.

Exclusion Criteria:

* Metastasis to the brain, problems during surgery leading to myocardial infarction or hemorrhage, cerebral infarction or hemorrhage, respiratory failure, non-healing surgical wound.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change of the score of the Trial Outcome Index (TOI) | Baseline to up to 12 weeks
  To measure health related quality of life (HRQOL), the TOI will be used,sum of the scores on the Lung Cancer Subscales (LCS) and the physical well-being and functional well-being subscales of the Functional Assessment of Cancer Therapy - Lung (FACT-L) scale. Frequencies, means and standard deviations of the patient characteristics will be compared between groups at baseline to assess the success of the randomization, and whether any baseline values need to be controlled for in analysis. Differences between groups in the change in outcome scores on the FACT-L, LSC, and TOI will be assessed using analysis of covariance, where covariates will include the stratification variable as well as any variables found to differ between groups at baseline.
Measures of pulmonary function | Baseline to up to 12 weeks
  Objective pulmonary function will be measured on a 3 measure spirometer ((FVC), forced expiratory volume in 1 second (FEV1) and peak expiratory flow rate (PEFR)). Since there are 3 measures of pulmonary function, the two groups will be compared using mixed model methods.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Shall, PT, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No